CLINICAL TRIAL: NCT00329472
Title: Randomized Phase III Trial of Neoadjuvant Chemotherapy Followed by Surgery Plus Adjuvant Chemotherapy Versus Surgery Plus Adjuvant Chemotherapy in Stage IB, IIA, IIB and T3N1 Non-small Cell Lung Cancer (ICON)
Brief Title: Efficacy Study of Induction Chemotherapy Before Surgery in Operable Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Samsung Medical Center (Other)
Responsible Party: Keunchil Park/Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-09-027
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

ARMS (2):
- Gem/Cis (Experimental): neoadjuvant chemotherapy: gemcitabine 1250mg/m2 D1,D8 & cisplatin 70mg/m2 , 2 cycles
  Interventions: Drug: gemcitabine, cisplatin
- no neoadjuvant chemotherapy (No Intervention)

INTERVENTIONS:
Drug: gemcitabine, cisplatin
  Arms: Gem/Cis

SUMMARY:
This study is randomized phase III trial designed to assess whether (preoperative) neoadjuvant chemotherapy followed by surgery plus adjuvant chemotherapy with gemcitabine and cisplatin (experimental treatment) improves 3-year disease-free survival, compared to surgery plus adjuvant chemotherapy with gemcitabine and cisplatin (standard treatment) in stage IB, IIA, IIB and T3N1 non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven NSCLC patients
* All patients must have:Clinical stage IB, IIA, IIB and T3N1 by mediastinoscopy, Chest CT and PET-CT
* 18 year of ages or older
* ECOG performance status 0-1
* Uni-dimensionally measurable lesion by RECIST criteria
* No prior chemotherapy or radiotherapy for NSCLC
* Pre-operative FEV1 ≥ 2.0 L evaluated within 28 days
* Adequate bone marrow function: Hb > 9.0 g/dL, WBC ≥ 4,000/μL, platelet count ≥ 100,000/μL
* Adequate liver and renal function: Total bilirubin < 2 x ULN, AST/ALT < 3 x ULN, serum creatinine ≤ 1.5 mg/dL, creatinine clearance ≥ 60 mL/min
* Written informed consent

Exclusion Criteria:

* Superior sulcus tumor
* Prior malignancy except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer at least 5 years
* Uncontrolled systemic illness such as DM, CHF, unstable angina or arrhythmia
* Recent myocardial infarction within 6 months
* Patients with post-obstructive pneumonia or serious infection
* Pregnant or nursing women (Women of reproductive potential have to agree to use an effective contraceptive method.)
* Patients with psychological problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival

SECONDARY OUTCOMES:
overall survival
pattern of relapse
quality of life
operative mortality and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Keunchil Park, M.D., Principal Investigator — Samsung Medical Center